CLINICAL TRIAL: NCT06401564
Title: Improving Functional and Cognitive Outcomes After Ischemic Stroke Using Virtual Reality Based Rehabilitation
Brief Title: Virtual Reality Based Rehabilitation After Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Good Samaritan Hospital (Unknown)
Responsible Party: Principal Investigator, Jason Mathew, Assistant Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2021-00237
Record Dates: First submitted 2024-04-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Stroke
Keywords: virtual reality; stroke rehabilitation; quality of life; upper extremity
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Therapy (Experimental)
  Interventions: Device: Virtual Reality Therapy

INTERVENTIONS:
Device: Virtual Reality Therapy — Each participant will receive one or two 20 minute VR sessions during their admission. Participants are able to pause or discontinue at any time. During each VR session, participants will use the REAL Immersive VR system and be equipped with a VR headset and 6 sensors attached to the torso, waist, and upper extremities. Patient will then undergo various virtual challenges guided by the physical or occupational therapist facilitating movements of the upper extremity, core, head, and neck.

SUMMARY:
Use the template below as a guide to write a brief study description in plain language. Tailor the text that appears in brackets and yellow to your research study. To finalize, delete the text in italics.

The goal of this single-arm study is to explore the use of early virtual reality-based rehabilitation as an adjunct to conventional physical/occupational therapy in adult patients with acute ischemic stroke. The main question it aims to answer is:

Feasibility and tolerability of using immersive Virtual Reality technology-based therapy for patients suffering from acute ischemic stroke in an inpatient hospital setting Participants will receive 1 or 2 virtual reality therapy sessions and complete surveys at the end of each session.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* MRI or CT imaging confirmed ischemic stroke
* Able to follow multistep commands

Exclusion Criteria:

* Plegia in both arms
* Previous reported history of vertigo or inner ear dysfunction
* Patients with epilepsy
* Patients who cannot begin therapy during admission
* Patients who are pregnant
* Patients with a pre-existing condition that interferes with virtual reality usage (e.g., visual impairment, limitation of either upper extremity or neck).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility survey | After each session up to 5 weeks
  The User Satisfaction Evaluation Questionnaire (USEQ) is a 14-item questionnaire evaluating satisfaction on a scale from 1 (not at all) to 5 (severely).
Simulator sickness questionnaire | After each session up to 5 weeks
  An evaluation tool for assessing the subjective severity of simulator sickness symptoms. A 16-item questionnaire evaluating different symptoms on a scale from 0 (not at all) to 4 (severe).

SECONDARY OUTCOMES:
Adverse events | After each session up to 5 weeks
  Frequency of adverse events such as dizziness, lightheadedness, nausea, headache, falls, fatigue, or other symptoms prompting program termination prior to end of a single 20-minute session
NIHSS | Hospital discharge, an average of 7 days
  NIHSS is a standardized method that uses a 42-point scale to measure the level of impairment caused by a stroke. The 42-point scale measures several aspects of brain function, including consciousness, vision, sensation, movement, speech, and language (0 = no stroke and 42 = severe stroke).
Modified Rankin Scale (mRS) | Hospital discharge, an average of 7 days
  The mRS incorporates mental as well as physical adaptations to the neurological deficits. It measures independence rather than performance of specific tasks. The mRS includes 15 items and takes approximately six minutes to complete. Scales consists of seven grades, from zero to six, with zero corresponding to no symptoms and six corresponding to death.
Duration of sessions | After each session up to 1 week
  Actual time spent using the Virtual Reality (VR) system
Time spent by therapist | After each session up to 1 week
  Time spent by therapist assisting patient including set-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Mathew, DO, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No